CLINICAL TRIAL: NCT01661036
Title: Cognitive Testing of the Family Life, Activity, Sun, Health, and Eating (FLASHE) Survey
Brief Title: Testing the FLASHE Survey
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912176; 12-C-N176
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-08-07

CONDITIONS: Cognitive Testing; Interview; Survey
Keywords: Cognitive Testing; Survey; Interview

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- The Family Life, Activity, Sun, Health, and Eating (FLASHE) Survey is designed to look at health-related topics. It is being developed for the Department of Health and Human Services. Researchers want to see how easy or difficult the FLASHE survey questions are to understand and answer. They will interview parents and teenagers to test the survey questions.

Objectives:

- To test the FLASHE survey questions on teenagers and their parents.

Eligibility:

* Adolescents between 11 and 18 years of age.
* Parents of the participating adolescents.

Design:

* Participants will have a one-on-one interview to test the survey questions. The interview will last up to an hour and a half. Participants will be allowed to skip any questions that they do not wish to answer.
* Participants will receive financial compensation for their time.

DETAILED DESCRIPTION:
The National Cancer Institute s (NCI) Division of Cancer Control and Population Sciences (DCCPS), Behavioral Research Program (BRP) proposes conducting formative research as an integral part of the development of a new data collection instrument, the Family Life, Activity, Sun, Health, and Eating (FLASHE) survey. Specifically, NCI proposes conducting cognitive testing with the objective of identifying potential sources of measurement or response errors within the questionnaires. Many of the questions are new questions that have not been previously tested, or previously-used questions that have never been used with a teenage population.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

The DCCPS contractor, Westat, will be conducting the study. Participants for the cognitive interviews will be recruited from the general population, and will include dyads of a parent or caregiver, and his/her teenage child between the ages of 11 and 18. Neither the contractor who will be coordinating the research (Westat) or NCI employees will be eligible to participate in the cognitive interviews. Westat will recruit respondents using a variety of methods including use of Westat s current database of potential participants and advertising on CraigsList in the local DC area under the Jobs postings within the subheading Et Cetera. Westat's digital media team will reach out to 100 local DC area (including lower Pennsylvania) publishers such as mommy and papi bloggers, health websites, giveaway publishers, and Facebook and Twitter users.

Ages: 11 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07-23; Study Completion 2015-08-07

PRIMARY OUTCOMES:
Survey Development | At time of interview

CONTACTS AND LOCATIONS:
Overall Officials: Linda C Nebeling, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States